CLINICAL TRIAL: NCT06340880
Title: Serratus Anterior Plane Block: Ultrasound Guided Versus Anatomical Landmark, A Randomized Control, Non-Inferiority Trial
Brief Title: Serratus Anterior Plane Block, Ultrasound vs Anatomical Landmark Guided.
Status: Completed | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Wesameldin Abelrahman Soltan, Associate Professor, Menoufia University
Other Study IDs: SAPB
Record Dates: First submitted 2024-03-24; First posted 2024-04-02 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Serratus Anterior Plane Block
Keywords: serratus anterior block; gynecomastia; anatomical landmark
MeSH Terms: conditions — Gynecomastia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ultrasound vs anatomical landmark SAPB: Forty subjects presenting for gynecomastia surgery will receive ultrasound guided block in one side (US group) and landmark guided block in the other side (LM group) with the same volume (25) ml and concentration (0.25 %) of bupivacaine.
  Interventions: Other: Serratus anterior plane block

INTERVENTIONS:
Other: Serratus anterior plane block — ultrasound guided SAPB vs anatomical landmark guided SAPB

SUMMARY:
This prospective, double-blinded randomized controlled trial aims to compare the efficacy of the serratus anterior plane block (SAPB) ultrasound guided versus anatomical landmark guided for gynecomastia surgery. And to detect if the anatomical landmark technique is inferior or not to the ultrasound guided technique. We hypothesize that anatomical landmark guided SAPB is not inferior to ultrasound guided SAPB.

DETAILED DESCRIPTION:
Gynecomastia means enlarged male breast. Minimally invasive liposuction and surgical intervention are possible remedies for such cases. Postoperative pain can be controlled by opioids or regional blocks like serratus anterior plane block. Ultrasound guided blocks are associated with high success rate; however, anatomical landmark guided blocks may give similar results. Our hypothesis was that landmark guided serratus anterior plane block would be non-inferior to ultrasound plane block. Subjects presenting for gynecomastia surgery will receive ultrasound guided block in one side (US group) and landmark guided block in the other side (LM group) with the same volume (25) ml and concentration (0.25 %) of bupivacaine. The primary outcome will be visual analogue score. Secondary outcomes include patient satisfaction and incidence of complications like pneumothorax. It will be carried out over 40 male patients, aged from (18 - 60) year-old, with ASA I or II classes who will undergo elective gynecomastia surgery. Patient with BMI ≥ 35, history of previous chest surgery, drug abuse, allergy to local anesthetics, psychiatric problems or patient refusal will be excluded from participation

ELIGIBILITY:
Inclusion Criteria:

* male patients, aged from (18 - 60) year-old, with ASA I or II classes who will undergo elective gynecomastia surgery

Exclusion Criteria:

* Patient with BMI ≥ 35, history of previous chest surgery, drug abuse, allergy to local anesthetics, psychiatric problems or patient refusal will be excluded from participation.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: male patients with gynecomastia
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
visual analouge score (VAS) | the first hour, postoperative
  11 point scale, 0 means no pain, 10 means worst pain.

SECONDARY OUTCOMES:
first call of analgesia | in the first 24 hours
  the time for the first call of analgesia
incidence of complications | in the first 24 hours
  pneumothorax, skin bruises
patient satisfaction | in the first 24 hours
  1-5 score, 1 means very dissatisfied, 5 means very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Wesamelsin A Soltan, MD, Principal Investigator — Menoufia University
Locations (1):
- Menoufia University Hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol can be shared with other researchers after finishing the research.
Supporting Information: Study Protocol
Time Frame: 2-3 months and will be available forever